CLINICAL TRIAL: NCT02859636
Title: Pronostic Value of Endothelial Dysfunction in Heart Failure
Acronym: Pro-ICARD
Status: Terminated | Type: Observational
Why Stopped: Not enough inclusions
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: P/2012/140
Record Dates: First submitted 2016-08-02; First posted 2016-08-09 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-08

CONDITIONS: Heart Decompensation; Cardiac Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum samples, endothelial progenitors
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The main objective is to evaluate the pronostic value of endothelial dysfonction in acute heart failure on a combined criteria associating cardiovascular mortality, nex hospitalisation for decompensated heart failure, cardiac graft or ventricular assistance 2 month and 1 year before acute heart failure.

ELIGIBILITY:
Inclusion Criteria:

* patients hospitalized for acute heart fialure with Left Ventricular Ejection Fraction (LVEF) < 45 % on echocardiography

Exclusion Criteria:

* Informed consent form not signed
* Cardiogenic, septic or hemorragic shock
* Acute coronary syndrom with elevated troponin
* valvular surgery or aorto-coronary graft during next 3 months
* Cancer
* Pregnancy
* life expectancy over than 1 year
* chronic renal impairment

Ages: 18 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with more than 18 years and less than 81 years, hospitalized for acute heart failure with left ventricular impairment (LVEF < 45%)
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2012-10; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
MR Proadrenomedulline | 6 months
catecholamins | 6 months
(untitled outcome) | 6 months
late endothelial progenitors | 6 months
Peripheral tissular perfusion | 6 months
  Near infra-red spectroscopy
mortality | 6 months
hospitalisation | 6 months